CLINICAL TRIAL: NCT04299958
Title: Observational Prospective Study on the Presence of Typical Migraine Features in Nummular Headache Patients: The Numamig Study
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, David García Azorín, Principal investigator, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI 20-1638
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Nummular Headache; Migraine; Headache Disorders, Primary
Keywords: Nummular headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient diary — In the first visit they will be examined by a neurologist with experience in headache disorders and NH diagnosis will be reviewed. Patients will be invited to participate into the study and they will provide and sign informed consent form. They will be instructed and trained to complete the prospective headache diary during 14 days. A follow up visit will be done within 15 to 30 days to review the data and analyze possible sources of bias.

SUMMARY:
Observational analytic study with prospective cohort design that aim to describe the presence of typical features of migraine in a cohort of nummular headache patients. The aim of the study is to analyze family history, epidemiology, clinical description, presence of prodromes, postdromes and response to treatment.

DETAILED DESCRIPTION:
Background:

Nummular headache (NH) is a primary headache included in the International Classification of Headache Disorders (ICHD) characterized by a well delimited superficial pain, with sharp border, felt in a rounded or elliptical 1-6 centimeters area. Pain might be continuous or intermittent. The key feature of nummular headache is the fixed superficial topography.

The real nature of this condition is still a matter of controversial. Some authors defend it as a specific condition with a particular pathophysiology; whereas others consider that it might be a localized form of migraine with a shared phenotype and pathophysiology.

Among the arguments that defend its existence as a differentiated entity we include: the older age of onset, the fixed and localized pain without pain in other territories, presence of trophic changes, the localized abnormality in pressure pain threshold determination, the description of secondary cases, the description of posttraumatic cases or the specific therapeutic response.

On the other hand, in some cases hypersensitivity to stimuli has been described, other typical migrainous symptoms such as nausea or vomiting might be present, and some patients respond to triptans or other migraine prophylactics.

Information is scarce about the presence of prodromes, postdromes or family history of migraine. Moreover, little is known about NH pathophysiology, some studies suggest an impairment in superficial sensory fibers because a localized alteration of pressure-pain threshold. No imaging or laboratory studies have been done so far.

This is a proof of concept study. The aim is to analyze if patients with a definite NH diagnosis according to ICHD present any shared epidemiological, clinical or therapeutical features with migraine.

Hypothesis:

Nummular headache might be a specific condition or it might share migraine biologic features. The detailed description of it might help to clarify whether if NH is a single entity or a focal presentation form of migraine.

Objective:

To describe the presence of typical features of migraine in a cohort of NH patients, including family history, epidemiology, clinical description, presence of prodromes or postdromes and response to treatment.

Methods:

The study has an observational analytic design following the Strengthening the Reporting of Observational in Epidemiology (STROBE) guidelines. Patients with definite nummular headache diagnosis according to The International Classification of Headache Disorders1 will be invited to participate. The study will be conducted in the Headache Unit of Hospital Clinico Universitario de Valladolid, a third level hospital sited in Valladolid, with a reference population of 280.000 people.

Intervention:

The study will be divided into different sections:

1. Family history of headache and in particular, migraine.
2. Epidemiology of NH patients.
3. Clinical phenotype and pattern of the headache.
4. Associated symptoms, presence of prodromes and postdromes.
5. Physical examination.
6. Prior treatment use, tolerability and response.

Selection of participants:

Recruitment will be recruited by a non-probabilistic sampling method by convenience and by formal invitation if they are included in the clinical registry of the Headache Unit of the Hospital Clinico Universitario de Valladolid.

In the first visit participants will be examined by a neurologist with experience in headache disorders and NH diagnosis will be reviewed. Patients will be invited to participate into the study and they will provide and sign informed consent form. They will be instructed and trained to complete the prospective headache diary during 14 days. A follow up visit will be done within 15 to 30 days to review the data and analyze possible sources of bias.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Nummular Headache (NH) according to the International Classification of Headache Disorders, 3rd version (ICHD-3).
2. More than 3 months of NH evolution.
3. No better accounted for by another ICHD-3 diagnosis.
4. Older than 18 years.
5. Capable of prospectively register headache characteristics in a diary.
6. Ability to provide informed consent form.

Exclusion Criteria:

1. Other primary or secondary headache, except for infrequent tension-type headache or medication overuse headache.
2. Major psychiatric disorders.
3. Alcoholism or drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite diagnosis of nummular headache that visit the headache outpatient clinic of Valladolid University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Family history of migraine | Through study completion, an average of 1 month
  To assess family history of migraine headache in nummular patients. We will build family tree up to 3 generations and we will ask patients to complete it by questioning their relatives.
Epidemiological pattern | Through study completion, an average of 1 month
  To determine age of onset, age when they were diagnosed, temporal pattern and frequency of headache.
Clinical phenotype | Through study completion, an average of 1 month
  To assess the clinical characteristics of nummular headache, analyzing the presence of typical features of migraine. Patients will complete a prospective headache diary for 15 days.
Presence of associated symptoms | Through study completion, an average of 1 month
  To assess the presence of symptoms such as nausea, vomiting, dizziness during the headache episodes.
Presence of prodromes | Through study completion, an average of 1 month
  To assess the presence of typical migraine prodromes before the headache episodes.
Presence of postdromes | Through study completion, an average of 1 month
  To assess the presence of typical migraine postdromes after the headache episode.
Presence of sensory disturbances | Through study completion, an average of 1 month
  To evaluate the presence of sensory changes such as hypoesthesia, hyperalgesia or allodinia upon examination.
Response to acute treatment | Through study completion, an average of 1 month
  To describe response to prior acute medications.
Response to prophylactic treatment | Through study completion, an average of 1 month
  To assess response to prior prophylactic treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
To be decided if anonymous data-sheets are available for other researchers upon reasonable request.

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Pareja JA, Caminero AB, Serra J, Barriga FJ, Baron M, Dobato JL, Vela L, Sanchez del Rio M. Numular headache: a coin-shaped cephalgia. Neurology. 2002 Jun 11;58(11):1678-9. doi: 10.1212/wnl.58.11.1678. PMID 12058099
- [Background] Trigo J, Garcia-Azorin D, Martinez Pias E, Sierra A, Chavarria A, Guerrero AL. Clinical characteristics of nummular headache and differentiation between spontaneous and posttraumatic variant: an observational study. J Headache Pain. 2019 Apr 8;20(1):34. doi: 10.1186/s10194-019-0981-4. PMID 30961529
- [Background] Garcia-Azorin D, Trigo-Lopez J, Sierra A, Blanco-Garcia L, Martinez-Pias E, Martinez B, Talavera B, Guerrero AL. Observational, open-label, non-randomized study on the efficacy of onabotulinumtoxinA in the treatment of nummular headache: The pre-numabot study. Cephalalgia. 2019 Dec;39(14):1818-1826. doi: 10.1177/0333102419863023. Epub 2019 Jul 4. PMID 31272194
- [Background] Cuadrado ML, Lopez-Ruiz P, Guerrero AL. Nummular headache: an update and future prospects. Expert Rev Neurother. 2018 Jan;18(1):9-19. doi: 10.1080/14737175.2018.1401925. Epub 2017 Nov 9. PMID 29103335